CLINICAL TRIAL: NCT01271543
Title: Comparing Hemodynamic Changes for Intubation With Shikani Intubating Stylet and Macintosh Laryngoscope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sonia Vaida, M.D, Vice Chair for Reasearch, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 35113; IRB protocol 35113 (Other: IRB protocol 35113)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia
Keywords: Comparison of hemodynamic; endotracheal intubation; changes induced by; performed; the aid of the SOS; as compared to the Macintosh Laryngoscope
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MacIntosh group (Active Comparator)
  Interventions: Device: Endotracheal Intubation
- Shikani optical stylet (Experimental)
  Interventions: Device: Endotracheal Intubation

INTERVENTIONS:
Device: Endotracheal Intubation — General anesthesia will be induced with fentanyl 1-2 mcg/kg, 2-3 mg/kg propofol and maintained with 50% air /50% oxygen and isoflurane. Neuromuscular blockade will be obtained with rocuronium 0.5 mg/kg. Laryngoscopy will be performed with Shikani optical stylet (SOS) (one size) or MacIntosh laryngoscope blade size 3 for women and size 4 for men. Endotracheal intubation will be performed with an endotracheal tube of internal diameter of 7.0 mm l for female patients and 8 mm for male in both groups. Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation. The patients will be questioned post-operatively about symptoms of a sore throat, hoarseness, dysphonia or dysphagia in the Post Anesthesia Care Unit and again 24 hours after surgery.

SUMMARY:
Because of its simplicity of function and reliability, direct laryngoscopy it is routinely used for endotracheal intubation during general anesthesia. However, direct laryngoscopy is fraught with concerns for cardiovascular stimulation during induction of general anesthesia. This can be attributed to the placement of the laryngoscope blade into the vallecula and then applying force in an upward direction to expose the glottic opening. The average force necessary for visualization of the glottic opening is approximately 5.4kg. This can lead to significant pressor responses and tachycardia though stimuli to supraglottic region.

An alternative airway management device is the Shikani optical stylet (SOS). It is an effective, safe and reusable intubation device that has been shown to be effective in cases of difficult intubation. It consists of a fiberoptic bundle within a J - shaped malleable stainless steel sheath. At the proximal end of the sheath is an eyepiece with an attachment to a light source. An adjustable "tube stop" firmly affixes the endotracheal tube to the stylet, and has a port to be able to deliver oxygen. (4) The operator inserts the tip of the stylet with the loaded endotracheal tube into the patient's oropharynx and under direct visualization through the eyepiece, is able to visualize the vocal cords. Because the end of the stylet is at the end of the endotracheal tube, it can be directly visualized to be entering trachea past the vocal cords.

The investigators hypothesize that endotracheal intubation performed by the aid of SOS by minimizing oropharyngolaryngeal stimulation will result in fewer hemodynamic changes in patients with normal airways as compared with the MacIntosh laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years, ASA I and II, normotensive, Mallampati class: I and II, thyromental distance > than 6.5 cm, interincisor distance > than 3 cm, BMI < 35 Kg/m2

Exclusion Criteria:

* Exclusion criteria: pregnant patients, known or expected difficult airway, gastroesophageal reflux, esophageal pathology, pulmonary pathology, cardiovascular pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PennState Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at Penn State Milton S. Hershey Medical Center
Pre-assignment Details: No events
Groups:
- MacIntosh Group: Endotracheal Intubation : General anesthesia will be induced with fentanyl 1-2 mcg/kg, 2-3 mg/kg propofol and maintained with 50% air /50% oxygen and isoflurane. Neuromuscular blockade will be obtained with rocuronium 0.5 mg/kg. Laryngoscopy will be performed with MacIntosh laryngoscope blade size 3 for women and size 4 for men. Endotracheal intubation will be performed with an endotracheal tube of internal diameter of 7.0 mm l for female patients and 8 mm for males. Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation. The patients will be questioned post-operatively about symptoms of a sore throat, hoarseness, dysphonia or dysphagia in the Post Anesthesia Care Unit and again 24 hours after surgery.
- Shikani Optical Stylet: Endotracheal Intubation : General anesthesia will be induced with fentanyl 1-2 mcg/kg, 2-3 mg/kg propofol and maintained with 50% air /50% oxygen and isoflurane. Neuromuscular blockade will be obtained with rocuronium 0.5 mg/kg. Laryngoscopy will be performed with Shikani optical stylet (SOS) (one size). Endotracheal intubation will be performed with an endotracheal tube of internal diameter of 7.0 mm l for female patients and 8 mm for males. Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation. The patients will be questioned post-operatively about symptoms of a sore throat, hoarseness, dysphonia or dysphagia in the Post Anesthesia Care Unit and again 24 hours after surgery.
Period: Overall Study
Arm/Group | MacIntosh Group | Shikani Optical Stylet
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Sample size of 30 patient for each group was calculated based on previous publications (2,3) to obtain of power of 80% and alfa of 0.05 to detect a 20 bpm for heart rate and 20 mmHg for blood pressure difference for paired hemodynamic data.
Groups:
- MacIntosh Group: Endotracheal Intubation : General anesthesia will be induced with fentanyl 1-2 mcg/kg, 2-3 mg/kg propofol and maintained with 50% air /50% oxygen and isoflurane. Neuromuscular blockade will be obtained with rocuronium 0.5 mg/kg. Laryngoscopy will be performed with a MacIntosh laryngoscope blade size 3 for women and size 4 for men. Endotracheal intubation will be performed with an endotracheal tube of internal diameter of 7.0 mm l for female patients and 8 mm for males. Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation. The patients will be questioned post-operatively about symptoms of a sore throat, hoarseness, dysphonia or dysphagia in the Post Anesthesia Care Unit and again 24 hours after surgery.
- Total: Total of all reporting groups
Arm/Group | MacIntosh Group | Shikani Optical Stylet | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 29 | 29
  >=65 years | 30 | 1 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11) | 39.6 (13) | 39.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate and Blood Pressure Double Product
Description: The double product was measured. The double product is calculated by multiplying the heart rate with the systolic blood pressure. It is also known as the rate pressure product and it is used to measure hemodynamic response.The double product is calculated from the values obtained preinduction, during intubation and after intubation.(5 minutes after intubation)The double products from each time point are averaged to get one mean double product value.
Time Frame: Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation.
Population: double product (DP) of systolic blood pressure multiplied by heart rate
Measure: Mean (Standard Deviation); unit: (beats/minute)*mmHg
Groups:
- Shikani Optical Stylet: Endotracheal Intubation : General anesthesia will be induced with fentanyl 1-2 mcg/kg, 2-3 mg/kg propofol and maintained with 50% air /50% oxygen and isoflurane. Neuromuscular blockade will be obtained with rocuronium 0.5 mg/kg. Laryngoscopy will be performed with a Shikani optical stylet (SOS) (one size). Endotracheal intubation will be performed with an endotracheal tube of internal diameter of 7.0 mm l for female patients and 8 mm for males. Noninvasive blood pressure and heart rate will be recorded preinduction, preintubation, and every min for the first 5 min after successful intubation. The patients will be questioned post-operatively about symptoms of a sore throat, hoarseness, dysphonia or dysphagia in the Post Anesthesia Care Unit and again 24 hours after surgery.
Arm/Group | MacIntosh Group | Shikani Optical Stylet
Number analyzed (Participants) | 29 | 29
(beats/minute)*mmHg | 9114 (1125) | 8804 (610)

2. Secondary Outcome: Time to Complete Laryngoscopy and Successful Intubation
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | MacIntosh Group | Shikani Optical Stylet
Number analyzed (Participants) | 29 | 29
seconds | 28.8 (14) | 37.41 (12)

ADVERSE EVENTS:
Arm/Group | MacIntosh Group | Shikani Optical Stylet
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
NO adverse events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No